CLINICAL TRIAL: NCT02992366
Title: IMMEDIATE IMPLANT PLACEMENT IN THE ESTHETIC ZONE: SOCKET SHIELD TECHNIQUE VERSUS EMPTY SOCKET TECHNIQUE FOR PRESERVATION OF LABIAL ALVEOLAR BONE INTEGRITY
Brief Title: : SOCKET SHIELD TECHNIQUE VERSUS EMPTY SOCKET TECHNIQUE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Khater Ali, Oral and Maxillofacial surgery resident in ministry of health, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairoshi-con
Record Dates: First submitted 2016-12-10; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Dental Implant Placement; Socket Shield Technique Implant Placement
Keywords: socket shield; volumetric tissue alteration; immediate implant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- socket shield (A) (Experimental): 1. Following local anesthetic infiltration opposite to the root to be extracted the root is sectioned in a mesiodistal direction along its long axis as far apical as possible.
  2. After sectioning the root into labial and palatal halves, the palatal half is removed with preservation of the labial root section.
  3. The labial half is prepared to be Flushing or 1mm above the labial alveolar crest. Then thinned slightly to a concave contour in an apico-coronal and mesiodistal direction.
  4. The implant will be inserted in place of the palatal half with the labial surface of the implant facing the labial root shield (root-implant interface)
  primary closure will not be attempted as the patients will undergo immediate non-functioning provisionization.
  Interventions: Procedure: implant placement
- conventional immediate implant (B) (Active Comparator): 1. Following local anesthetic infiltration opposite to the root to be extracted non traumatic extraction of the tooth or remaining root by periotome.
  2. The implant fixture will be inserted in the empty socket by conventional manner.
  primary closure will not be attempted as the patients will undergo immediate non-functioning provisionization.
  Interventions: Procedure: implant placement

INTERVENTIONS:
Procedure: implant placement — implant placement

SUMMARY:
To evaluate the clinical and radiographic outcomes of socket shield technique compared with conventional immediate implant placement.

DETAILED DESCRIPTION:
To evaluate the clinical and radiographic outcomes of socket shield technique compared with conventional immediate implant placement.

PICO

* P: patient require immediate dental implant placement for esthetic consideration
* I: socket shield technique
* C: conventional immediate implant placement
* O:

Outcome name Measuring device Measuring unit Primary outcome Vertical and horizontal bone level Cone beam Computer Tomography (CBCT) Millimeter Secondary outcome (a) Pocket probing depth Periodontal probe Millimeter Secondary outcome (b) Labial Alveolar crestal bone height compared with the lingual side Cone beam Computer Tomography (CBCT) Millimeter

ELIGIBILITY:
Inclusion Criteria:

1. Patients with remaining roots in the esthetic zone with intact periodontal condition indicated for extraction.
2. Physically able to tolerate conventional surgical and restorative procedures
3. Signing of an informed consent form
4. Implant insertion torque > 32 N cm with good primary stability

Exclusion Criteria:

1. Systemic diseases contraindicating implant placement eg uncontrolled diabetes
2. Severe bruxism
3. Active infection in the teeth to be treated
4. Vertical root fractures with displacement in the teeth of the surgical area

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Vertical and horizontal bone level | 9 months

SECONDARY OUTCOMES:
Pocket probing depth | 9 months
Labial Alveolar crestal bone height compared with the lingual side | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Galal G. Beheiri, professor, Study Director — senior supervisor

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cardaropoli G, Araujo M, Lindhe J. Dynamics of bone tissue formation in tooth extraction sites. An experimental study in dogs. J Clin Periodontol. 2003 Sep;30(9):809-18. doi: 10.1034/j.1600-051x.2003.00366.x. PMID 12956657
- [Background] Araujo MG, Sukekava F, Wennstrom JL, Lindhe J. Ridge alterations following implant placement in fresh extraction sockets: an experimental study in the dog. J Clin Periodontol. 2005 Jun;32(6):645-52. doi: 10.1111/j.1600-051X.2005.00726.x. PMID 15882225
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Background] Buser D, Martin W, Belser UC. Optimizing esthetics for implant restorations in the anterior maxilla: anatomic and surgical considerations. Int J Oral Maxillofac Implants. 2004;19 Suppl:43-61. PMID 15635945
- [Background] Botticelli D, Persson LG, Lindhe J, Berglundh T. Bone tissue formation adjacent to implants placed in fresh extraction sockets: an experimental study in dogs. Clin Oral Implants Res. 2006 Aug;17(4):351-8. doi: 10.1111/j.1600-0501.2006.01270.x. PMID 16907764
- [Background] Fickl S, Zuhr O, Wachtel H, Bolz W, Huerzeler MB. Hard tissue alterations after socket preservation: an experimental study in the beagle dog. Clin Oral Implants Res. 2008 Nov;19(11):1111-8. doi: 10.1111/j.1600-0501.2008.01575.x. PMID 18983313
- [Background] AMLER MH, JOHNSON PL, SALMAN I. Histological and histochemical investigation of human alveolar socket healing in undisturbed extraction wounds. J Am Dent Assoc. 1960 Jul;61:32-44. doi: 10.14219/jada.archive.1960.0152. No abstract available. PMID 13793201
- [Background] Fickl S, Zuhr O, Wachtel H, Stappert CF, Stein JM, Hurzeler MB. Dimensional changes of the alveolar ridge contour after different socket preservation techniques. J Clin Periodontol. 2008 Oct;35(10):906-13. doi: 10.1111/j.1600-051X.2008.01305.x. Epub 2008 Aug 17. PMID 18713258
- [Background] Pietrokovski J, Massler M. Alveolar ridge resorption following tooth extraction. J Prosthet Dent. 1967 Jan;17(1):21-7. doi: 10.1016/0022-3913(67)90046-7. No abstract available. PMID 5224784
- [Background] Lang NP, Pun L, Lau KY, Li KY, Wong MC. A systematic review on survival and success rates of implants placed immediately into fresh extraction sockets after at least 1 year. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:39-66. doi: 10.1111/j.1600-0501.2011.02372.x. PMID 22211305
- [Background] Botticelli D, Berglundh T, Lindhe J. Hard-tissue alterations following immediate implant placement in extraction sites. J Clin Periodontol. 2004 Oct;31(10):820-8. doi: 10.1111/j.1600-051X.2004.00565.x. PMID 15367183
- [Background] Hammerle CH, Araujo MG, Simion M; Osteology Consensus Group 2011. Evidence-based knowledge on the biology and treatment of extraction sockets. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:80-2. doi: 10.1111/j.1600-0501.2011.02370.x. PMID 22211307
- [Background] Chen ST, Wilson TG Jr, Hammerle CH. Immediate or early placement of implants following tooth extraction: review of biologic basis, clinical procedures, and outcomes. Int J Oral Maxillofac Implants. 2004;19 Suppl:12-25. PMID 15635942
- [Background] Fickl S, Schneider D, Zuhr O, Hinze M, Ender A, Jung RE, Hurzeler MB. Dimensional changes of the ridge contour after socket preservation and buccal overbuilding: an animal study. J Clin Periodontol. 2009 May;36(5):442-8. doi: 10.1111/j.1600-051X.2009.01381.x. PMID 19419446
- [Background] Vermylen K, Collaert B, Linden U, Bjorn AL, De Bruyn H. Patient satisfaction and quality of single-tooth restorations. Clin Oral Implants Res. 2003 Feb;14(1):119-24. doi: 10.1034/j.1600-0501.2003.140116.x. PMID 12562374
- [Background] Baumer D, Zuhr O, Rebele S, Schneider D, Schupbach P, Hurzeler M. The socket-shield technique: first histological, clinical, and volumetrical observations after separation of the buccal tooth segment - a pilot study. Clin Implant Dent Relat Res. 2015 Feb;17(1):71-82. doi: 10.1111/cid.12076. Epub 2013 Apr 30. PMID 23631704
- [Background] Cherel F, Etienne D. Papilla preservation between two implants: a modified socket-shield technique to maintain the scalloped anatomy? A case report. Quintessence Int. 2014 Jan;45(1):23-30. doi: 10.3290/j.qi.a30765. PMID 24392492
- [Background] Kan JY, Rungcharassaeng K. Proximal socket shield for interimplant papilla preservation in the esthetic zone. Int J Periodontics Restorative Dent. 2013 Jan-Feb;33(1):e24-31. doi: 10.11607/prd.1346. PMID 23342355
- [Background] Scheuber S, Bosshardt D, Bragger U, von Arx T. [Implant therapy following trauma of the anterior teeth - a new method for alveolar ridge preservation after post-traumatic ankylosis and external root resorption]. Schweiz Monatsschr Zahnmed. 2013;123(5):417-39. French, German. PMID 23720038
- [Background] Parlar A, Bosshardt DD, Unsal B, Cetiner D, Haytac C, Lang NP. New formation of periodontal tissues around titanium implants in a novel dentin chamber model. Clin Oral Implants Res. 2005 Jun;16(3):259-67. doi: 10.1111/j.1600-0501.2005.01123.x. PMID 15877745
- [Background] Davarpanah M, Szmukler-Moncler S. Unconventional implant treatment: I. Implant placement in contact with ankylosed root fragments. A series of five case reports. Clin Oral Implants Res. 2009 Aug;20(8):851-6. doi: 10.1111/j.1600-0501.2008.01653.x. PMID 19604282
- [Background] Donos N, Mardas N, Chadha V. Clinical outcomes of implants following lateral bone augmentation: systematic assessment of available options (barrier membranes, bone grafts, split osteotomy). J Clin Periodontol. 2008 Sep;35(8 Suppl):173-202. doi: 10.1111/j.1600-051X.2008.01269.x. PMID 18724850
- [Background] Salama M, Ishikawa T, Salama H, Funato A, Garber D. Advantages of the root submergence technique for pontic site development in esthetic implant therapy. Int J Periodontics Restorative Dent. 2007 Dec;27(6):521-7. PMID 18092446
- [Background] Bowers GM, Chadroff B, Carnevale R, Mellonig J, Corio R, Emerson J, Stevens M, Romberg E. Histologic evaluation of new attachment apparatus formation in humans. Part III. J Periodontol. 1989 Dec;60(12):683-93. doi: 10.1902/jop.1989.60.12.683. PMID 2614633
- [Background] Hurzeler MB, Zuhr O, Schupbach P, Rebele SF, Emmanouilidis N, Fickl S. The socket-shield technique: a proof-of-principle report. J Clin Periodontol. 2010 Sep;37(9):855-62. doi: 10.1111/j.1600-051X.2010.01595.x. PMID 20712701
- [Background] Chen ST, Buser D. Esthetic outcomes following immediate and early implant placement in the anterior maxilla--a systematic review. Int J Oral Maxillofac Implants. 2014;29 Suppl:186-215. doi: 10.11607/jomi.2014suppl.g3.3. PMID 24660198